CLINICAL TRIAL: NCT05105828
Title: Predictive Power of Share Wave Fibro Scan in HCC After HCV Infection
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Roshdy Elkhayat, Principle investigator, Assiut University
Other Study IDs: Share wave fibro scan in HCC
Record Dates: First submitted 2021-10-23; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post Hepatitis C patients with hepatocellular carcinoma: post Hepatitis C patients with hepatocellular carcinoma above 18 years
  Interventions: Diagnostic Test: Share wave fibro scan
- control group: post Hepatitis C patients without hepatocellular carcinoma above 18 years
  Interventions: Diagnostic Test: Share wave fibro scan

INTERVENTIONS:
Diagnostic Test: Share wave fibro scan — Shear wave elastography (SWE) measures LS by quantifying the velocity of shear waves produced in the liver tissue and uses a normal B-mode ultrasound probe for measuring LS in real time. In addition, SWE imaging using the Aixplorer system provides a high frame-rate and may be able to provide more accurate scoring of fibrosis

SUMMARY:
Shear wave electrography score allows stratification of HCC risk in a noninvasive and reliable way and can guide the surveillance strategy for HCC in patients with CLD

DETAILED DESCRIPTION:
Liver fibrosis is common to all chronic liver disease (CLD) , With time, this progressive disruption of hepatic architecture can develop into cirrhosis, characterized by "diffuse conversion of normal liver architecture into structurally abnormal nodules", About1% to 4% of patients with HCV-induced liver cirrhosis are diagnosed with HCC each year .

The historical gold standard for quantifying fibrosis is liver biopsy, but its invasive nature and potential for complications make it unpopular among patients and impractical for serial assessments of CLD. Furthermore, since histological lesions are not uniformly distributed across the liver parenchyma, this allows for large sampling error. The need for credible alternatives to biopsy has stimulated research into non-invasive methods of fibrosis assessment, including serum biomarkers , axial imaging and transient elastography.

FibroScan™ (Echosens, Paris, France) allows a non-invasive liver stiffness measurement (LSM), it is a relatively simple, highly reproducible and operator independent technique which examines an area 100 times that of a biopsy, reducing sampling bias , Shear wave elastography (SWE) measures LS by quantifying the velocity of shear waves produced in the liver tissue and uses a normal B-mode ultrasound probe for measuring LS in real time. In addition, SWE imaging using the Aixplorer system provides a high frame-rate and may be able to provide more accurate scoring of fibrosis .

ELIGIBILITY:
Inclusion Criteria:

* Post hepatitis C with HCC

Exclusion Criteria:

* hepatic encephalopathy, ascites or pregnancy, hepatorenal syndrome or hepato-pulmonary syndrome, right side heart failure (liver congestion), extra hepatic tumors, history of liver transplantation, cholestasis, and hepatitis B patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Post hepatitis C with HCC above 18 years
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Shear wave elastography score | through study completion, an average of 1 year
  it measures liver stiffness as it is a rapid technique taking less than 5 min that can be easily performed at bedside or in outpatient clinic,according to the manufacturer's recommendations and the machine scale result ranges from 2.5 to 75 kPa with normal value around 5.5 kPa

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Tsochatzis EA, Bosch J, Burroughs AK. Liver cirrhosis. Lancet. 2014 May 17;383(9930):1749-61. doi: 10.1016/S0140-6736(14)60121-5. Epub 2014 Jan 28. PMID 24480518
- [Background] Sumida Y, Nakajima A, Itoh Y. Limitations of liver biopsy and non-invasive diagnostic tests for the diagnosis of nonalcoholic fatty liver disease/nonalcoholic steatohepatitis. World J Gastroenterol. 2014 Jan 14;20(2):475-85. doi: 10.3748/wjg.v20.i2.475. PMID 24574716
- [Background] Taylor-Robinson SD. Applications of magnetic resonance spectroscopy to chronic liver disease. Clin Med (Lond). 2001 Jan-Feb;1(1):54-60. doi: 10.7861/clinmedicine.1-1-54. PMID 11358078
- [Background] Ferraioli G, Tinelli C, Dal Bello B, Zicchetti M, Filice G, Filice C; Liver Fibrosis Study Group. Accuracy of real-time shear wave elastography for assessing liver fibrosis in chronic hepatitis C: a pilot study. Hepatology. 2012 Dec;56(6):2125-33. doi: 10.1002/hep.25936. Epub 2012 Aug 31. PMID 22767302